CLINICAL TRIAL: NCT01602549
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Dose Ranging Study to Assess the Effect of Repeat Doses of GSK962040 on the Pharmacokinetics of L-DOPA in Subjects With Parkinson's Disease Exhibiting Delayed Gastric Emptying
Brief Title: A Study to Assess the Effect of Repeat Doses of GSK962040 on the Pharmacokinetics of L-DOPA in Subjects With Parkinson's Disease Exhibiting Delayed Gastric Emptying
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 115816
Record Dates: First submitted 2012-05-17; First posted 2012-05-21 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — N-(3-fluorophenyl)-1-((4-(((3S)-3-methyl-1-piperazinyl)methyl)phenyl)acetyl)-4-piperidinamine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort (Experimental): 1:2 ratio, placebo, 50 mg administered orally once daily for 7-9 days
  Interventions: Drug: GSK962040 (25 mg tablet); Drug: Placebo

INTERVENTIONS:
Drug: GSK962040 (25 mg tablet) — 25 mg tablet
Drug: Placebo — matching placebo tablet

SUMMARY:
Gastric emptying is the end-result of a complex and carefully regulated series of events which follow the ingestion of a meal, each of which is dependent on the other and subject to neurohormonal control. Motilin is an endogenous peptide, produced mainly in the duodenum, whose physiological action is mediated by motilin receptors located on enteric neurons, peripheral terminals of the vagus, and on the smooth muscle of the gut. Motilin and non-peptide agonists at motilin receptors increases the gastric emptying rate and therefore provide a potential approach to the treatment of a range of clinical conditions in which delayed gastric emptying is thought to be part of the physiopathology and may be contributory to symptoms. Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by degeneration of nigrostriatal dopaminergic neurones. It affects 1.5% of the global population over 65 years of age. Cardinal symptoms comprise bradykinesia, rigidity, resting tremors and postural instability. Gastrointestinal dysfunction, including gastroparesis, is a frequent feature of PD affecting approximately 90% of patients, and is caused by autonomic dysfunction as well as an adverse effect of antiparkinsonian drug therapy. The therapeutic mainstay for PD treatment is the neutral amino acid L-3,4-dihydroxyphenylalanine (L-DOPA), a dopamine prodrug, as it provides the most rapid and effective symptomatic control of motor impairment in PD. The primary determinant of L-DOPA bioavailability is gastric emptying (GE); delays in GE slow delivery of L-DOPA to its proximal small intestinal absorption sites, increasing the extent of presystemic metabolism, and leading to slowed and diminished absorption.

DETAILED DESCRIPTION:
MOT115816 will be conducted as a multi-center, randomized, double-blind, placebo controlled study to investigate the ability of the motilin receptor agonist GSK962040 to improve L-DOPA pharmacokinetics (PK) by enhancing gastric emptying via motilin receptor agonism. Subjects will be randomized to receive 50 mg GSK962040 or placebo in a 2:1 ratio administered orally once daily for 7-9 days. The study will consist of a screening/baseline period, a treatment period, and a 14-day post treatment safety follow-up visit. During this period participants will be asked to attend the study center for 5 visits 3 of which will last approximately 5 hours. The duration of each patient's participation in the study from screening to follow-up visit will be approximately 7-8 weeks. For three of the visits, subjects will visit the clinical unit fasted and prior to taking their first morning L-DOPA dose. Volunteers will undergo a complete physical (including cardiovascular monitoring (ECG), vital signs, blood samples, and medical history), measurement of plasma L-DOPA levels, completion of patient diary to capture the amount of awake time (in hours) spent "on" without dyskinesias, "on" with troublesome dyskinesias, "on" with non-troublesome dyskinesias, and "off" and gastric symptoms, non-motor and motor symptoms assessments (MDS-UPDRS rating scale and "finger taps") and measurement of gastric emptying rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease (according to modified Hoehn & Yahr criteria Stages II-IV) and with suboptimal motor control on L-DOPA or L-DOPA combination therapy (i.e. wearing off, peak dose dyskinesias, delayed on or no-on effects)
* Subjects receiving a stable regimen of L-DOPA for at least four weeks prior to screening
* Patient has gastric half-time of emptying > or = 70 min as determined by 13C oral breath test
* Between 40 and 80 years of age, inclusive.
* Patient has never had a gastrectomy, nor major gastric surgical procedure or any evidence of bowel obstruction or strictures within the previous 12 months
* Dosage of any concomitant medications has been stable for at least 4 weeks
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Child-bearing potential and is abstinent or agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until at least 5 days post-last dose.
* ALT < 2xULN; alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single or Average QTc, QTcB or QTcF< 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* Late stage advanced subjects with incapacitating peak dose or biphasic dyskinesia ona stable L-DOPA regime.
* Presence, or history within the previous 3 months, of significant and/or uncontrolled psychiatric, neurological (other than Parkinson's disease), gastro-intestinal, hematological, endocrinologic, neurological (other than Parkinson's disease), cardiovascular disease, active malignancy (other than basal cell cancer) or other condition that would in the opinion of the investigator or medical monitor make the subject unsuitable for inclusion in this clinical study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Patient has a gastric pacemaker
* Patient is on chronic enteral (e.g., feeding tube) or parenteral feeding
* Patient has evidence of severe cardiovascular autonomic neuropathy (e.g. history of recurrent syncope in the last 6 months)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unable to refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until followup.
* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study (e.g., prokinetic drugs, macrolide antibiotics (erythromycin), GLP-1 mimetics)
* Unable to refrain from use of prohibited medications listed in Section 9 within the restricted timeframe relative to the first dose of study medication.
* The patient has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day time-period.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- GSK Investigational Site, Randwick, New South Wales, Australia
- Germany (6):
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Jena, Thuringia
- GSK Investigational Site, Uppsala, Sweden
- United Kingdom (3):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Norwich

REFERENCES:
- [Derived] Marrinan SL, Otiker T, Vasist LS, Gibson RA, Sarai BK, Barton ME, Richards DB, Hellstrom PM, Nyholm D, Dukes GE, Burn DJ. A randomized, double-blind, placebo-controlled trial of camicinal in Parkinson's disease. Mov Disord. 2018 Feb;33(2):329-332. doi: 10.1002/mds.27259. Epub 2017 Dec 26. PMID 29278279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a Screening/Baseline Period, a Treatment Period, and a 14-day post-treatment safety Follow-up Visit. Participants were randomized to receive GSK962040 50 milligrams or placebo in a 2:1 ratio; one participant was randomized to receive GSK962040 125 mg.
Groups:
- Placebo: Participants received placebo administered orally once daily for 7 to 9 days.
- GSK962040 Total: Participants received GSK962040 50 milligrams (mg) (except for one participant who received GSK962040 125 mg) administered orally once daily for 7 to 9 days.
Period: Overall Study
Arm/Group | Placebo | GSK962040 Total
Started | 19 | 38
Completed | 18 | 37
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The GSK962040 data include 37 subjects who received the 50-mg dose and 1 subject who received the 125-mg dose" in the baseline description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK962040 Total | Total
Number analyzed (Participants) | 19 | 38 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (8.04) | 67.4 (7.97) | 67.1 (7.93)
Gender [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 29 | 37
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 19 | 38 | 57

OUTCOME MEASURES:

1. Primary Outcome: Dose-normalized Levodopa (L-DOPA) Area Under the Plasma Concentration-time Curve From Zero to 4 Hours AUC(0-4) at Baseline
Description: Dose-normalized L-DOPA AUC(0-4) was derived from L-DOPA plasma concentration-time data. AUC is a measure of levodopa exposure.
Time Frame: Baseline
Population: Pharmacodynamic (PD)/Efficacy Population: participants receiving >=1 dose placebo/GSK962040 50 mg. Only those participants available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour/milliliter/milligram
Groups:
- GSK962040 50 mg: Participants received GSK962040 50 milligrams (mg) administered orally once daily for 7 to 9 days.
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 17 | 33
Nanograms*hour/milliliter/milligram | 24.13 (37.5) | 24.81 (36.1)

2. Primary Outcome: Dose-normalized L-DOPA AUC(0-4) at Day 1 and Day 8
Description: Dose-normalized L-DOPA AUC(0-4) was derived from L-DOPA plasma concentration-time data. The adjusted means and ratios (GSK962040 50 mg: Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit, Baseline L-dopa pharmacokinetic (PK) parameter, and Baseline gastric emptying half-time as fixed effects, and participant as a random effect. AUC is a measure of levodopa exposure
Time Frame: Day 1 and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms*hour/milliliter/milligram
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Nanograms*hour/milliliter/milligram
  Day 1, n=17, 31 | 26.6 (0.058) | 25.7 (0.047)
  Day 8, n=17, 32 | 27.1 (0.058) | 24.1 (0.047)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg : Placebo Day 1; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.965, 95% CI 2-sided [0.831 to 1.120] — Day 1: The adjusted means (AMs) and ratios were estimated using a mixed model (MM) fitting treatment, visit, treatment*visit, Baseline L-dopa PK parameter and Baseline gastric emptying half time as fixed effects, and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg : Placebo Day 8; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.886, 95% CI 2-sided [0.763 to 1.029] — Day 8: The AMs and ratios were estimated using a mixed model fitting treatment, visit, treatment*visit, Baseline L-dopa PK parameter and Baseline gastric emptying half time as fixed effects, and participant as a random effect
Statistical Analysis 3: Comparison: GSK962040 50 mg; Day 8: Day 1; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.937, 95% CI 2-sided [0.850 to 1.033] — Day 8:Day 1: The AMs and ratios were estimated using a mixed model fitting treatment, visit, treatment*visit, Baseline L-dopa PK parameter and Baseline gastric emptying half time as fixed effects, and participant as a random effect
Statistical Analysis 4: Comparison: Placebo; Day 8:Day 1 Placebo; Test type: Superiority or Other; Ratio of adjusted geometric means = 1.020, 95% CI 2-sided [0.890 to 1.170] — [estimate comment as in outcome 2, analysis 3]

3. Primary Outcome: Dose-normalized L-DOPA Maximum Observed Concentration (Cmax) at Baseline
Description: Dose-normalized L-DOPA Cmax was derived from L-DOPA plasma concentration-time data.
Time Frame: Baseline
Population: PD/Efficacy Population. Only those participants available at the specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter/milligram
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 17 | 35
Nanograms/milliliter/milligram | 12.77 (28.0) | 12.89 (42.6)

4. Primary Outcome: Dose-normalized L-DOPA Cmax at Day 1 and Day 8
Description: Dose-normalized L-DOPA Cmax was derived from L-DOPA plasma concentration-time data. The adjusted means and ratios were estimated using a mixed model fitting treatment, visit, treatment*visit, Baseline L-dopa PK parameter, and Baseline gastric emptying half-time as fixed effects, and participant as a random effect.
Time Frame: Day 1 and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Nanograms/milliliter/milligram
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Nanograms/milliliter/milligram
  Day 1, n=18, 35 | 13.4 (0.081) | 11.6 (0.065)
  Day 8, n=17, 35 | 11.6 (0.083) | 11.8 (0.065)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.864, 95% CI 2-sided [0.702 to 1.064] — Day 1: The AMs and ratios were estimated using a mixed model fitting treatment, visit, treatment*visit, Baseline L-dopa PK parameter and Baseline gastric emptying half time as fixed effects, and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Ratio of adjusted geometric means = 1.018, 95% CI 2-sided [0.824 to 1.257] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: GSK962040 50 mg; Day 8 VS Day 1 GSK962040 50 mg; Test type: Superiority or Other; Ratio of adjusted geometric means = 1.018, 95% CI 2-sided [0.889 to 1.166] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Placebo; Day 8 Vs Day 1 Placebo; Test type: Superiority or Other; Ratio of adjusted geometric means = 0.865, 95% CI 2-sided [0.709 to 1.055] — [estimate comment as in outcome 2, analysis 3]

5. Primary Outcome: L-DOPA Time of Occurrence of Cmax (Tmax) at Baseline, Day 1,and Day 8
Description: L-DOPA Tmax was derived from L-DOPA plasma concentration-time data.
Time Frame: Baseline, Day 1, and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Hours
  Baseline, n=17, 35 | 1.50 [0.3 to 3.6] | 2.00 [0.3 to 4.0]
  Day 1, n=18, 35 | 1.61 [0.5 to 3.4] | 1.50 [0.3 to 3.5]
  Day 8, n=17, 35 | 2.00 [0.5 to 3.5] | 1.55 [0.3 to 4.0]
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; Day 1; Test type: Superiority or Other; p = 0.157, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; Day 8; Test type: Superiority or Other; p = 0.186, Wilcoxon rank-sum test

6. Primary Outcome: L-DOPA Terminal Phase Half-life (t1/2) at Baseline, Day 1, and Day 8
Description: L-DOPA t1/2 was derived from L-DOPA plasma concentration-time data. This endpoint was not assessed because there were insufficient L-DOPA data/profiles to calculate this parameter.
Time Frame: Baseline, Day 1, and Day 8
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Gastric Half Emptying Time (GE t1/2) at Baseline (BL), Day 1, and Day 8
Description: Gastric half emptying time is the time taken for half the contents of the stomach to empty. Gastric emptying was measured using the 13C-oral breath test, which is a tracer method that utilizes 13C, a non-radioactive isotope. Basal breath samples were obtained after an overnight fast or otherwise after 4 hours of fasting following a light meal. On Day 1 and Day 8, participants were then dosed with GSK962040 and additional breath test samples were taken prior to administration of a 13C-labelled test meal. The test meal was consumed approximately 80 minutes later. After consumption of the test meal, breath samples were collected at pre-specified time points over an approximately 4 hour period following the test meal. For the duration of the breath test, no food or drink were allowed. The 13C breath content was determined by isotope ratio mass spectrometry. GE t1/2 was determined by using the cumulative percentage of the administered dose of 13C excreted in breath over 4 hours.
Time Frame: Baseline, Day 1, and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Minutes
  Baseline, n=19, 37 | 99.6 (21.26) | 96.9 (21.67)
  Day 1, n=19, 37 | 97.5 (15.81) | 91.9 (21.47)
  Day 8, n=17, 36 | 98.7 (25.03) | 90.6 (26.75)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -4.239, 95% CI 2-sided [-16.015 to 7.537] — Day 1: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit, and Baseline gastric half emptying time as fixed effects, and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -5.327, 95% CI 2-sided [-17.567 to 6.914] — Day 8: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit, and Baseline gastric half emptying time as fixed effects, and participant as a random effect

8. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Scores at Baseline, Day 1, and Day 8 (Pre-levodopa Dose)
Description: The MDS-UPDRS is used to assess the status of Parkinson's Disease. It has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination), and Part IV (motor complications). Each part is made up of several questions, with each question given a score ranging from 0 (normal) to 4 (severe). Part I and Part II consist of 13 items each, and have a score ranging between 0 (normal) and 52 (severe). Part III consists of 33 items, and has a score ranging between 0 (normal) and 132 (severe). Part IV consists of 6 items, and has a score ranging between 0 (normal) and 24 (severe). The total score is the summed score of all four parts and ranges between 0 (normal) and 260 (severe). A higher score indicates more severe symptoms.
Time Frame: Baseline, Day 1, and Day 8 at pre-levodopa dose
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Scores on a scale
  Part I: Baseline, n=19, 37 | 9.1 (4.56) | 10.1 (6.17)
  Part I: Day 1, n=19, 37 | 10.1 (4.98) | 8.6 (5.12)
  Part I: Day 8, n=18, 36 | 10.0 (5.25) | 7.1 (4.67)
  Part II: Baseline, n=19, 37 | 14.9 (7.09) | 12.5 (6.33)
  Part II: Day 1, n=19, 37 | 16.1 (9.09) | 11.5 (6.54)
  Part II: Day 8, n=18, 36 | 15.3 (9.29) | 10.3 (6.37)
  Part III: Baseline, n=19, 37 | 42.2 (14.63) | 38.0 (18.95)
  Part III: Day 1, n=19, 37 | 40.4 (17.56) | 34.9 (17.97)
  Part III: Day 8, n=18, 36 | 44.2 (19.25) | 34.0 (17.46)
  Part IV: Baseline, n=19, 37 | 5.5 (2.70) | 5.3 (3.63)
  Part IV: Day 1, n=19, 37 | 5.9 (3.07) | 5.2 (3.61)
  Part IV: Day 8, n=18, 36 | 5.7 (3.79) | 4.5 (3.41)
  Total: Baseline, n=19, 37 | 71.7 (23.53) | 65.8 (27.02)
  Total: Day 1, n=19, 37 | 72.5 (29.01) | 60.2 (25.90)
  Total: Day 8, n=18, 36 | 75.2 (34.27) | 55.9 (25.34)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; Part I-GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -2.16, 95% CI [-3.90 to -0.41] — Day 1; Part I: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; Part I-GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -3.63, 95% CI 2-sided [-5.41 to -1.85] — Day 8; Part I: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 3: Comparison: Placebo vs GSK962040 50 mg; Part II- GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -2.29, 95% CI 2-sided [-4.65 to 0.07] — Day 1; Part II: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 4: Comparison: Placebo vs GSK962040 50 mg; Part II- GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -2.46, 95% CI 2-sided [-4.85 to -0.07] — Day 8; Part II: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 5: Comparison: Placebo vs GSK962040 50 mg; Part III -GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -5.38, 95% CI 2-sided [-10.28 to -0.49] — Day 8; Part III: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 6: Comparison: Placebo vs GSK962040 50 mg; Part IV-GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -0.56, 95% CI 2-sided [-1.65 to 0.54] — Day 1; Part IV: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 7: Comparison: Placebo vs GSK962040 50 mg; Part IV-GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -0.90, 95% CI 2-sided [-2.02 to 0.22] — Day 8; Part IV: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 8: Comparison: Placebo vs GSK962040 50 mg; Total- GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -6.69, 95% CI 2-sided [-13.77 to 0.39] — Day 1; Total: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 9: Comparison: Placebo vs GSK962040 50 mg; Total- GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -12.5, 95% CI 2-sided [-19.67 to -5.29] — Day 8; Total: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect
Statistical Analysis 10: Comparison: Placebo vs GSK962040 50 mg; Part III- GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -1.70, 95% CI 2-sided [-6.53 to 3.13] — Day 1; Part III: The AMs and differences (GSK 962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit interaction, and Baseline MDS-UPDR score as fixed effects, and participant as a random effect

9. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Scores at Baseline, Day 1, and Day 8 (Pre-dose; 120, 180, and 240 Minutes Post-dose)
Description: as for outcome 8
Time Frame: Baseline, Day 1, and Day 8 at pre-dose and 120, 180, and 240 minutes (min) post-dose (PD); Follow-up visit (up to Day 25)
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Scores on a scale
  Baseline, pre-dose, n=19, 37 | 42.2 (14.63) | 38.0 (18.95)
  Baseline, 120 minutes post-dose, n=19, 37 | 33.1 (16.61) | 27.7 (16.04)
  Baseline, 180 minutes post-dose, n=19, 36 | 30.3 (14.55) | 27.5 (14.21)
  Baseline, 240 minutes post-dose, n=19, 37 | 31.6 (16.27) | 29.2 (16.62)
  Day 1, pre-dose, n=19, 37 | 40.4 (17.56) | 34.9 (17.97)
  Day 1,120 minutes post-dose, n=19, 37 | 32.3 (15.01) | 26.2 (16.25)
  Day 1, 180 minutes post-dose, n=19, 37 | 31.0 (17.10) | 25.5 (18.04)
  Day 1, 240 minutes post-dose, n=19, 37 | 32.7 (20.50) | 27.2 (17.68)
  Day 8, pre-dose n=18, 36 | 44.2 (19.25) | 34.0 (17.46)
  Day 8, 120 minutes post-dose, n=18, 36 | 32.3 (14.90) | 24.2 (14.24)
  Day 8, 180 minutes post-dose, n=18, 36 | 33.3 (16.17) | 25.1 (14.27)
  Day 8, 240 minutes post-dose, n=18, 36 | 37.1 (20.19) | 25.4 (15.27)
  Follow-up, n=19, 37 | 30.3 (13.45) | 24.9 (11.79)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; Pre dose: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -3.14, 95% CI 2-sided [-9.07 to 2.78] — Day 1; Pre-dose: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; 120 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -3.18, 95% CI 2-sided [-9.11 to 2.75] — Day 1; 120 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 3: Comparison: Placebo vs GSK962040 50 mg; 180 min PD: GSK962040 50 mg Vs Placebo Day 1:; Test type: Superiority or Other; Difference in AMs of change from BL = -3.66, 95% CI 2-sided [-9.59 to 2.27] — Day 1; 180 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 4: Comparison: Placebo vs GSK962040 50 mg; 240 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -4.15, 95% CI 2-sided [-10.07 to 1.76] — Day 1; 240 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 5: Comparison: Placebo vs GSK962040 50 mg; Pre dose: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -6.80, 95% CI 2-sided [-12.79 to -0.81] — Day 8; Pre-dose: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 6: Comparison: Placebo vs GSK962040 50 mg; 120 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -3.97, 95% CI 2-sided [-9.96 to 2.03] — Day 8; 120 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 7: Comparison: Placebo vs GSK962040 50 mg; 180 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -5.29, 95% CI 2-sided [-11.29 to 0.71] — Day 8; 180 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect
Statistical Analysis 8: Comparison: Placebo vs GSK962040 50 mg; 240 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -8.90, 95% CI 2-sided [-14.88 to -2.91] — Day 8; 240 min PD: The AMs and differences (GSK962040 minus Placebo) were estimated using a mixed model fitting treatment, visit, treatment*visit*time point interaction, and Baseline UPDRS-3 score as fixed effects, and participant as a random effect

10. Secondary Outcome: Period Mean Amount of Hours Spent "ON," "ON" Without Dyskinesia, "ON" With Non-troublesome Dyskinesia, "ON" With Troublesome Dyskinesia, and "OFF" at Baseline and During the Treatment Period (Days 1-8), Week 1 of Follow-up, and Week 2 of Follow-up
Description: Participants were provided with the "ON/OFF" diary to capture details of the amount of awake time spent on/off of PD symptoms, and were asked to complete the diary daily. Participants checked the box most appropriate for their dominant motor state in the preceding 30-minute period. The catergories included: "ON" (including "ON without dyskinesia" and "ON with non-troublesome dyskinesia"), "ON" with troublesome dyskinesia (TD), and "OFF." For Baseline, data were collected for 2 days prior to Day 1, and the mean value of the 2 days was used.
Time Frame: Baseline, Days 1-8, Week 1 of Follow-up (Days 6 and 7 of Follow-up; up to Day 16), and Week 2 of Follow-up (Days 13 and 14 of Follow-up; up to Day 23)
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
hours
  Baseline: "ON," n=18, 37 | 11.21 (3.602) | 11.31 (3.021)
  Baseline: "ON" without dyskinesia, n=18, 37 | 10.11 (4.069) | 9.65 (3.787)
  Baseline: "ON" with non-TD, n=18, 37 | 1.10 (1.787) | 1.66 (2.956)
  Baseline: "ON" with TD, n=18, 37 | 0.54 (1.240) | 0.40 (1.292)
  Baseline: "OFF," n=18, 37 | 4.92 (3.417) | 4.23 (2.484)
  Treatment period: "ON," n=18, 36 | 10.61 (3.927) | 12.44 (3.375)
  Treatment period: "ON" without dyskinesia, n=18,36 | 9.82 (4.042) | 10.47 (4.479)
  Treatment period: "ON" with non-TD, n=18, 36 | 0.79 (1.875) | 1.98 (2.987)
  Treatment period: "ON" with TD, n=18, 36 | 0.47 (1.548) | 0.59 (1.985)
  Treatment period: "OFF," n=18, 36 | 5.57 (4.364) | 2.94 (2.954)
  Week 1 of FU: "ON," n=18, 36 | 11.00 (3.309) | 12.13 (3.134)
  Week 1 of FU: "ON" without dyskinesia, n=18, 36 | 10.17 (4.232) | 10.63 (3.948)
  Week 1 of FU: "ON" with non-TD, n=18, 36 | 0.83 (1.933) | 1.50 (2.369)
  Week 1 of FU: "ON" with TD, n=18, 36 | 0.71 (2.083) | 0.52 (1.986)
  Week 1 of FU: "OFF," n=18, 36 | 4.83 (3.700) | 3.31 (2.642)
  Week 2 of FU: "ON," n=16, 32 | 11.34 (3.580) | 11.69 (3.562)
  Week 2 of FU: "ON" without dyskinesia, n=16, 32 | 11.13 (4.138) | 9.98 (4.872)
  Week 2 of FU: "ON" with non-TD, n=16, 32 | 0.22 (0.875) | 1.70 (2.838)
  Week 2 of FU: "ON" with TD, n=16, 32 | 0.38 (1.500) | 0.80 (2.362)
  Week 2 of FU: "OFF," n=16, 32 | 4.47 (3.601) | 3.36 (2.857)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; OFF: Treatment Period; Test type: Superiority or Other; Difference in AMs of change from BL = -2.31, 95% CI 2-sided [-3.71 to -0.90] — OFF: Treatment Period: The AMs and differences (GSK962040 minus Placebo) were estimated using an analysis of covariance (ANCOVA) model fitting treatment and Baseline amount of hours spent ON/OFF as main effects
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; ON: Treatment Period; Test type: Superiority or Other; Difference in AMs of change from BL = 1.88, 95% CI 2-sided [0.28 to 3.48] — ON: Treatment Period: The AMs and differences (GSK962040 minus Placebo) were estimated using an analysis of covariance (ANCOVA) model fitting treatment and Baseline amount of hours spent ON/OFF as main effects

11. Secondary Outcome: Number of Times a Participant Could Alternatively Tap Two Counter Keys 30 Centimeters Apart in 1 Minute (Min) at Baseline, Day1, Day 8, and Follow-up
Description: Participants were asked to alternatively tap two keys 30 centimeters apart in 1 minute in two trials with the most affected hand or the dominant hand in symmetric disease. The finger tapping was scored manually by the study staff. The finger-tapping assessment was repeated at eight separate time points (pre-dose, 0 min, 30 min, 60 min, 90 min, 120 min, 180 min, and 240 min post-dose) at each visit (Baseline, Day 1, and Day 8). At each time point, the mean of the two assessments was calculated.
Time Frame: Baseline, Day 1, and Day 8 at pre-dose and 0, 30, 60, 90, 120, 180, and 240 minutes post-dose; Follow-up visit (up to Day 25)
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Finger taps per minute
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Finger taps per minute
  Baseline: pre-dose, n=19, 37 | 92.4 (47.53) | 77.8 (38.00)
  Baseline: 0 min, n=19, 35 | 91.2 (49.84) | 80.1 (35.28)
  Baseline: 30 min, n=19, 34 | 89.3 (42.91) | 85.2 (41.45)
  Baseline: 60 min, n=19, 36 | 88.6 (42.32) | 89.3 (45.32)
  Baseline: 90 min, n=19, 36 | 91.2 (44.14) | 90.8 (45.18)
  Baseline: 120 min, n=19, 37 | 92.6 (40.99) | 92.0 (43.37)
  Baseline: 180 min, n=19, 37 | 94.1 (47.19) | 92.8 (44.86)
  Baseline: 240 min, n=19, 37 | 95.2 (44.60) | 93.2 (46.17)
  Day 1: pre-dose, n=19, 36 | 92.3 (43.44) | 85.1 (40.05)
  Day 1: 0 min, n=19, 364 | 90.7 (40.78) | 86.8 (44.65)
  Day 1: 30 min, n=18, 35 | 93.4 (43.95) | 92.4 (49.92)
  Day 1: 60 min, n=18, 35 | 93.8 (44.80) | 94.6 (44.06)
  Day 1: 90 min, n=19, 34 | 97.7 (50.46) | 91.4 (42.09)
  Day 1: 120 min, n=19, 35 | 99.9 (50.51) | 96.4 (42.06)
  Day 1: 180 min, n=18, 36 | 99.0 (49.44) | 92.3 (41.01)
  Day 1: 240 min, n=18, 36 | 98.2 (51.97) | 97.6 (48.40)
  Day 8: pre-dose, n=18, 35 | 95.7 (40.90) | 92.8 (43.92)
  Day 8: 0 min, n=18, 35 | 92.0 (44.30) | 91.1 (42.90)
  Day 8: 30 min, n=18, 34 | 95.8 (45.07) | 92.2 (41.14)
  Day 8: 60 min, n=18, 35 | 94.6 (46.80) | 93.2 (39.01)
  Day 8: 90 min, n=18, 34 | 95.0 (48.82) | 95.5 (42.60)
  Day 8: 120 min, n=18, 35 | 97.2 (47.67) | 97.4 (42.34)
  Day 8: 180 min, n=18, 34 | 96.8 (52.50) | 101.2 (49.86)
  Day 8: 240 min, n=18, 35 | 98.3 (53.30) | 102.8 (51.84)
  Follow-up: n=18, 35 | 104.4 (48.13) | 105.7 (56.59)
Statistical Analysis 1: Comparison: Placebo vs GSK962040 50 mg; Pre-dose: Day GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -2.83, 95% CI 2-sided [-21.79 to 16.13] — Day 1, pre-dose: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 2: Comparison: Placebo vs GSK962040 50 mg; 0 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = 0.58, 95% CI 2-sided [-18.39 to 19.56] — Day 1, 0 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 3: Comparison: Placebo vs GSK962040 50 mg; Day 1, 30 min PD; Test type: Superiority or Other; Difference in AMs of change from BL = 1.84, 95% CI 2-sided [-17.18 to 20.86] — Day 1, 30 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 4: Comparison: Placebo vs GSK962040 50 mg; 60 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = 0.28, 95% CI 2-sided [-18.72 to 19.28] — Day 1, 60 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 5: Comparison: Placebo vs GSK962040 50 mg; 90 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -3.38, 95% CI 2-sided [-22.35 to 15.58] — Day 1, 90 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 6: Comparison: Placebo vs GSK962040 50 mg; 120 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -4.18, 95% CI 2-sided [-23.13 to 14.76] — Day 1, 120 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 7: Comparison: Placebo vs GSK962040 50 mg; 180 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = -6.39, 95% CI 2-sided [-25.36 to 12.58] — Day 1, 180 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 8: Comparison: Placebo vs GSK962040 50 mg; 240 min PD: GSK962040 50 mg Vs Placebo Day 1; Test type: Superiority or Other; Difference in AMs of change from BL = 0.77, 95% CI 2-sided [-18.20 to 19.75] — Day 1, 240 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 9: Comparison: Placebo vs GSK962040 50 mg; Pre-dose: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = 0.51, 95% CI 2-sided [-18.51 to 19.52] — Day 8, pre-dose: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 10: Comparison: Placebo vs GSK962040 50 mg; 0 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = 3.32, 95% CI 2-sided [-15.70 to 22.33] — Day 8, 0 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 11: Comparison: Placebo vs GSK962040 50 mg; 30 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -2.94, 95% CI 2-sided [-21.97 to 16.08] — Day 8, 30 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 12: Comparison: Placebo vs GSK962040 50 mg; 60 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -3.12, 95% CI 2-sided [-22.13 to 15.88] — Day 8, 60 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 13: Comparison: Placebo vs GSK962040 50 mg; 90 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -1.38, 95% CI 2-sided [-20.40 to 17.63] — Day 8, 90 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 14: Comparison: Placebo vs GSK962040 50 mg; 120 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = -0.71, 95% CI 2-sided [-19.70 to 18.28] — Day 8, 120 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 15: Comparison: Placebo vs GSK962040 50 mg; 180 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = 3.02, 95% CI 2-sided [-15.98 to 22.02] — Day 8, 180 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect
Statistical Analysis 16: Comparison: Placebo vs GSK962040 50 mg; 240 min PD: GSK962040 50 mg Vs Placebo Day 8; Test type: Superiority or Other; Difference in AMs of change from BL = 4.08, 95% CI 2-sided [-14.91 to 23.07] — Day 8, 240 min PD: The AMs/differences (GSK962040 minus Placebo) were estimated using a MM fitting treatment, visit, time point (TP), treatment*visit*TP interaction, and BL score as fixed effects, TP as a repeated effect, and par. as a random effect

12. Secondary Outcome: Total Daily L-DOPA Equivalent Dose at Baseline and on Days 1, 2, 3, 4, 5, 6, 7, 8, and 9
Description: Various formulations of L-DOPA were utilized by participants for the treatment of Parkinson's Disease. The total daily L-DOPA equivalent dose was calculated as the sum of all L-DOPA equivalent doses for each L-DOPA-containing drug taken on the same day.
Time Frame: Baseline and Days 1, 2, 3, 4, 5, 6, 7, 8, and 9
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 19 | 37
Milligrams
  Baseline, n=19, 37 | 113.2 (41.14) | 164.5 (119.66)
  Day 1, n=19, 37 | 353.9 (174.85) | 368.6 (216.54)
  Day 2, n=19, 36 | 465.8 (229.61) | 514.5 (300.44)
  Day 3, n=19, 36 | 481.6 (243.79) | 516.9 (299.98)
  Day 4, n=19, 36 | 481.6 (241.50) | 518.3 (313.07)
  Day 5, n=19, 36 | 484.2 (243.13) | 503.0 (293.48)
  Day 6, n=17, 36 | 516.2 (249.21) | 511.3 (307.31)
  Day 7, n=17, 35 | 486.8 (247.51) | 499.6 (310.57)
  Day 8, n=17, 34 | 191.2 (175.43) | 281.3 (234.00)
  Day 9, n=0, 5 | 0.0 (0.0) | 235.0 (121.96)

13. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Day 1 and Day 8
Description: Blood pressure measurements were taken at pre-dose and at 0 min (completion of meal) on Day 1 and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 1, and Day 8
Population: All Subjects Population (ASP): all participants who received >=1 dose of study medication. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Millimeters of mercury
  SBP, Day 1: 0 min, n=19, 37, 38 | -4.0 (12.05) | -2.5 (18.66) | -2.1 (18.58)
  SBP, Day 8: pre-dose, n=18, 36, 37 | -2.8 (13.24) | -3.9 (13.19) | -3.7 (13.06)
  SBP, Day 8: 0 min, n=18, 36, 37 | -3.4 (11.55) | -1.0 (15.04) | -1.1 (14.84)
  DBP, Day 1: 0 min, n=19, 37, 38 | -5.4 (7.67) | -0.9 (7.51) | -0.7 (7.55)
  DBP, Day 8: pre-dose, n=18, 36, 37 | -4.2 (6.88) | -0.9 (8.54) | -0.8 (8.48)
  DBP, Day 8: 0 min, n=18, 36, 37 | -3.7 (5.81) | 0.9 (8.32) | 0.9 (8.21)

14. Secondary Outcome: Change From Baseline in Heart Rate at Day 1 and Day 8
Description: Heart rate measurements were taken at pre-dose and 0 min (completion of meal) on Day 1 and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 1, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Beats per minute
  Day 1: 0 min, n=19, 37, 38 | -2.2 (7.30) | 0.8 (9.19) | 0.5 (9.26)
  Day 8: pre-dose, n=18, 36, 37 | -2.9 (7.67) | 0.6 (6.12) | 0.0 (6.84)
  Day 8: 0 min, n=18, 36, 37 | -2.5 (7.64) | -0.5 (6.80) | -0.5 (6.71)

15. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Findings at Day 1 and Day 8
Description: ECG measurements were taken at pre-dose and 0 min (completion of meal) on Day 1 and Day 8. The Baseline value was the Day 1 pre-dose value. ECG findings were categorized as normal, abnormal - not clinically significant, and abnormal - clinically significant (CS), based on interpretation by the site.
Time Frame: Day 1 and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Participants
  Day 1: pre-dose, Normal, n=19, 37, 38 | 14 | 17 | 18
  Day 1: pre-dose, Abnormal - Not CS, n=19, 37, 38 | 5 | 19 | 19
  Day 1: pre-dose, Abnormal - CS, n=19, 37, 38 | 0 | 1 | 1
  Day 1: 0 min, Normal, n=19, 37, 38 | 12 | 16 | 16
  Day 1: 0 min, Abnormal - Not CS, n=19, 37, 38 | 7 | 20 | 21
  Day 1: 0 min, Abnormal - CS, n=19, 37, 38 | 0 | 1 | 1
  Day 8: pre-dose, Normal, n=18, 36, 37 | 14 | 18 | 19
  Day 8: pre-dose, Abnormal - Not CS, n=18, 36, 37 | 4 | 17 | 17
  Day 8: pre-dose, Abnormal - CS, n=18, 36, 37 | 0 | 1 | 1
  Day 8: 0 min, Normal, n=18, 36, 37 | 12 | 19 | 20
  Day 8: 0 min, Abnormal - Not CS, n=18, 36, 37 | 6 | 16 | 16
  Day 8: 0 min, Abnormal - CS, n=18, 36, 37 | 0 | 1 | 1

16. Secondary Outcome: Change From Baseline in Albumin (ALB) and Total Protein (TP) at Day 4 and Day 8
Description: ALB and TP measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Grams per liter
  ALB, Day 4, n=18, 34, 35 | 0.06 (2.313) | -0.38 (2.155) | -0.37 (2.124)
  ALB, Day 8, n=18, 34, 35 | 0.11 (2.220) | -0.33 (2.084) | -0.29 (2.065)
  TP, Day 4, n=18, 30, 31 | -0.3 (3.28) | -0.9 (3.93) | -1.0 (3.97)
  TP, Day 8, n=15, 31, 32 | -0.0 (3.24) | -0.3 (3.72) | -0.3 (3.66)

17. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), and Gamma Glutamyl Transferase (GGT) at Day 4 and Day 8
Description: ALP, ALT, AST, and GGT measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
International units per liter
  ALP, Day 4, n=19, 33, 34 | -0.8 (5.26) | 2.4 (14.14) | 2.2 (13.98)
  ALP, Day 8, n=18, 34, 35 | -0.1 (7.66) | 1.4 (13.35) | 1.2 (13.21)
  ALT, Day 4, n=19, 33, 34 | -6.4 (10.45) | -5.9 (9.77) | -7.1 (11.72)
  ALT, Day 8, n=18, 34, 35 | -1.6 (6.88) | -0.4 (5.46) | -0.6 (5.57)
  AST, Day 4, n=19, 32, 33 | 0.2 (3.16) | -1.2 (2.89) | -1.3 (2.96)
  AST, Day 8, n=16, 31, 32 | 0.6 (4.55) | 1.0 (3.65) | 0.9 (3.63)
  GGT, Day 4, n=19, 33, 34 | -0.8 (3.20) | -0.8 (3.06) | -0.9 (3.04)
  GGT, Day 4, n=18, 33, 34 | -0.1 (5.22) | -1.0 (5.02) | -1.0 (4.95)

18. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide Content (CO2)/Bicarbonate (BC), Glucose, Potassium, Sodium, Urea/Blood Urea Nitrogen (BUN), and Uric Acid (UA) at Day 4 and Day 8
Description: Calcium, chloride, CO2/BC, glucose, potassium, sodium, urea/BUN, and UA measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Millimoles per liter
  Calcium, Day 4, n=19, 34, 35 | 0.010 (0.0746) | -0.009 (0.0659) | -0.011 (0.0667)
  Calcium, Day 8, n=18, 35, 36 | 0.026 (0.0756) | -0.018 (0.0662) | -0.017 (0.0652)
  Chloride, Day 4, n=19, 33, 34 | -1.37 (1.832) | -0.42 (2.346) | -0.41 (2.311)
  Chloride, Day 8, n=18, 33, 34 | 0.39 (2.570) | 0.52 (1.734) | 0.53 (1.710)
  CO2/BC, Day 4, n=9, 21, 22 | -0.06 (2.833) | 0.16 (2.602) | 0.20 (2.546)
  CO2/BC, Day 8, n=8, 22, 23 | 0.51 (2.053) | 0.23 (2.139) | 0.13 (2.141)
  Glucose, Day 4, n=19, 35, 36 | 1.14 (2.944) | 0.14 (1.198) | 0.15 (1.185)
  Glucose, Day 8, n=18, 36, 36 | -0.03 (0.865) | 0.09 (0.594) | -0.09 (0.594)
  Potassium, Day 4, n=19, 32, 33 | 0.008 (0.3393) | 0.168 (0.3408) | 0.151 (0.3497)
  Potassium, Day 8, n=16, 31, 32 | 0.055 (0.3405) | 0.048 (0.2897) | 0.043 (0.2862)
  Sodium, Day 4, n=19, 34, 35 | -0.89 (2.787) | -0.56 (1.779) | -0.51 (1.772)
  Sodium, Day 8, n=18, 34, 35 | 1.39 (3.202) | 0.21 (1.647) | 0.29 (1.690)
  Urea/BUN, Day 4, n=17, 32, 33 | -0.27 (1.757) | 0.00 (1.496) | -0.02 (1.477)
  Urea/BUN, Day 8, n=17, 34, 35 | -0.63 (1.318) | 0.13 (1.308) | 0.14 (1.289)
  UA, Day 4, n=16, 30, 31 | -14.22 (23.416) | 0.53 (29.735) | -0.78 (30.127)
  UA, Day 8, n=14, 29, 30 | -1.56 (22.601) | 6.39 (30.819) | 6.17 (30.306)

19. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Absolute Neutrophil Count (ANC), and Platelet Count (PC) at Day 4 and Day 8
Description: Basophils, eosinophils, lymphocytes, monocytes, total ANC, and PC measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Giga (10^9) cells per liter
  Basophils, Day 4, n=19, 34, 35 | -0.003 (0.0200) | -0.006 (0.0247) | -0.006 (0.0244)
  Basophils, Day 8, n=17, 35, 36 | -0.006 (0.0153) | -0.001 (0.0195) | -0.001 (0.0192)
  Eosinophils, Day 4, n=19, 34, 35 | 0.003 (0.1219) | -0.031 (0.0584) | -0.034 (0.0599)
  Eosinophils, Day 8, n=17, 35, 36 | -0.016 (0.0519) | -0.001 (0.0466) | 0.000 (0.0467)
  Lymphocytes, Day 4, n=19, 34, 35 | 0.093 (0.4326) | 0.044 (0.3592) | 0.033 (0.3592)
  Lymphocytes, Day 8, n=17, 35, 36 | -0.049 (0.3258) | 0.076 (0.5874) | 0.073 (0.5793)
  Monocytes, Day 4, n=19, 34, 35 | 0.006 (0.1313) | 0.002 (0.0923) | 0.004 (0.0913)
  Monocytes, Day 8, n=17, 35, 36 | -0.004 (0.0860) | -0.013 (0.0928) | -0.013 (0.0916)
  Total ANC , Day 4, n=19, 34, 35 | 0.021 (0.8866) | 0.392 (0.9480) | 0.406 (0.9377)
  Total ANC , Day 8, n=17, 35, 36 | 0.007 (0.8586) | -0.114 (0.8500) | -0.122 (0.8392)
  PC, Day 4, n=19, 34, 35 | 4.5 (18.45) | 3.6 (18.76) | 3.3 (18.53)
  PC, Day 8, n=17, 35, 36 | 1.8 (24.42) | 1.4 (22.97) | 0.7 (22.97)

20. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC) at Day 4 and Day 8
Description: Hemoglobin and MCHC measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Grams per liter
  Hemoglobin, Day 4, n=19, 34, 35 | -2.3 (6.53) | -2.0 (6.35) | -2.3 (6.44)
  Hemoglobin, Day 8, n=17, 35, 36 | -2.4 (4.27) | -2.3 (4.71) | -2.2 (4.64)
  MCHC, Day 4, n=13, 24, 24 | -0.0 (8.85) | 0.6 (8.83) | 0.6 (8.83)
  MCHC, Day 8, n=12, 25, 25 | 0.4 (8.30) | -2.3 (8.47) | -2.3 (8.47)

21. Secondary Outcome: Change From Baseline in Hematocrit at Day 4 and Day 8
Description: Hematocrit measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: proportion of 1
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
proportion of 1
  Day 4, n=19, 34, 35 | -0.0059 (0.02331) | -0.0059 (0.02029) | -0.0067 (0.02051)
  Day 8, n=17, 35, 36 | -0.0044 (0.01383) | -0.0037 (0.01702) | -0.0039 (0.01682)

22. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) at Day 4 and Day 8
Description: MCH measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Picograms
  Day 4, n=19, 34, 35 | -0.12 (0.464) | -0.06 (0.744) | 0.07 (0.737)
  Day 8, n=17, 35, 36 | 0.03 (0.718) | -0.20 (0.832) | 0.19 (0.826)

23. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) at Day 4 and Day 8
Description: MCV measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Femtoliters
  Day 4, n=19, 34, 35 | -0.13 (1.945) | -0.14 (1.339) | -0.17 (1.334)
  Day 8, n=17, 35, 36 | 0.72 (1.322) | -0.05 (1.401) | -0.06 (1.381)

24. Secondary Outcome: Change From Baseline in Red Blood Cell Count (RBC) and White Blood Cell Count (WBC) at Day 4 and Day 8
Description: RBC and WBC measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Giga (10^9) cells per liter
  RBC, Day 4, n=19, 34, 35 | -0.055 (0.2345) | 0.068 (0.2138) | -0.074 (0.2140)
  RBC, Day 8, n=17, 35, 36 | -0.073 (0.1270) | 0.041 (0.1752) | -0.043 (0.1730)
  WBC, Day 4, n=19, 34, 35 | 0.140 (0.9284) | 0.390 (1.0592) | 0.392 (1.0437)
  WBC, Day 8, n=17, 35, 36 | -0.036 (0.8961) | -0.154 (0.9006) | -0.161 (0.8886)

25. Secondary Outcome: Change From Baseline in Reticulocytes (RET) at Day 4 and Day 8
Description: RET measurements were taken at pre-dose on Day 1 (Baseline), Day 4, and Day 8. The Baseline value was the Day 1 pre-dose value. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline value.
Time Frame: Baseline, Day 4, and Day 8
Population: ASP. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Mean (Standard Deviation); unit: Tera (10^12) cells per liter
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Tera (10^12) cells per liter
  RET, Day 4, n=16, 28, 29 | 0.000 (0.0075) | 0.002 (0.0093) | 0.001 (0.0098)
  RET, Day 8, n=13, 28, 29 | 0.004 (0.0080) | 0.001 (0.0093) | 0.001 (0.0095)

26. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect, is associated with liver injury and impaired liver function, or are serious events as per the medical or scientific judgment.
Time Frame: From the start of study medication until Follow-up (up to Day 25)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 Total
Number analyzed (Participants) | 19 | 37 | 38
Participants
  Any AE | 17 | 23 | 24
  Any SAE | 2 | 2 | 2

27. Secondary Outcome: GSK962040 Area Under the Plasma Concentration-time Curve From Zero to 5.5 Hours (AUC[0-5.5] and Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC[0-inf]) at Days 1 and 8
Description: GSK AUC(0-5.5) and AUC(0-inf) were derived from GSK962040 plasma concentration-time data. Only participants who received GSK962040 50 mg were analyzed. AUC is a measure of levodopa exposure. Data for AUC(0-inf) was analyzed and was only available for Day 1 and not for Day 8.
Time Frame: Day 1 and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms.hour/milliliter
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 0 | 36
Nanograms.hour/milliliter
  AUC(0-5.5): Day 1 |  | 1632.5 (38.1)
  AUC(0-5.5): Day 8 |  | 3036.9 (45.8)
  AUC(0-inf): Day 1 |  | 2972.8 (49.2)

28. Secondary Outcome: GSK962040 Percentage of AUC(0-inf) Obtained by Extrapolation (%AUCex) at Day 1
Description: GSK962040 %AUCex was derived from GSK962040 plasma concentration-time data. %AUCex is the percentage of the AUC(0-inf) extrapolated from the last PK sample drawn to infinity. This parameter is only reported in conjunction with single-dose AUC(0-inf). Only participants who received GSK962040 50 mg were analyzed. AUC is a measure of levodopa exposure.
Time Frame: Day 1
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 0 | 36
Percentage |  | 41.64 (28.9)

29. Secondary Outcome: GSK962040 Cmax at Day1 and Day 8
Description: GSK962040 Cmax was derived from GSK962040 plasma concentration-time data. Only participants who received GSK962040 50 mg were analyzed.
Time Frame: Day 1 and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 0 | 36
Nanograms/milliliter
  Day 1 |  | 501.0 (45.4)
  Day 8 |  | 788.3 (46.0)

30. Secondary Outcome: GSK962040 Tmax at Day1 and Day 8
Description: GSK962040 tmax was derived from GSK962040 plasma concentration-time data. Only participants who received GSK962040 50 mg were analyzed.
Time Frame: Day 1 and Day 8
Population: PD/Efficacy Population. Participants with available data (n=X, X in category titles) were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Placebo | GSK962040 50 mg
Number analyzed (Participants) | 0 | 36
Hours
  Day 1 |  | 0.750 [0.25 to 3.50]
  Day 8 |  | 1.000 [0.25 to 3.72]

ADVERSE EVENTS:
Time Frame: Post-randomization adverse events include those that occured on or after the randomization date.
Groups:
- GSK962040 125 mg: Participants received GSK962040 125 milligrams (mg) administered orally once daily for 7 to 9 days.
Arm/Group | Placebo | GSK962040 50 mg | GSK962040 125 mg
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/37 | 0/1
Other Adverse Events (participants affected / at risk) | 17/19 | 21/37 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | GSK962040 50 mg (N=37) | GSK962040 125 mg (N=1)
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | GSK962040 50 mg (N=37) | GSK962040 125 mg (N=1)
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 5 | 0
Chills (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 9 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0
Clumsiness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Metamorphopsia (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Micturition disorder (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.